CLINICAL TRIAL: NCT02895087
Title: Circadian HIV RNA Oscillations and Outcomes of Stress
Brief Title: Study to Explore Natural Daily Variation and Impact of Stress in HIV Levels
Acronym: CHRONOS
Status: Completed | Type: Observational
Sponsor: University of Melbourne (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: U19AI096109 (NIH)
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV
Keywords: diurnal variation; stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Part 1: Diurnal Variation cohort (total 15 participants) - no longer recruiting Blood samples
  Part 2: Stress cohort (total 20 participants) - no longer recruiting Blood samples Saliva Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Diurnal Variation Group: Cohort recruitment - open to recruitment
  Interventions: Other: Diurnal Variation Group
- Cohort 2: External Stress Group: Cohort recruitment - closed to recruitment
  Interventions: Other: External Stress Group

INTERVENTIONS:
Other: Diurnal Variation Group — This intervention occurs over one 24-hour period. Eligible participants will be required to be admitted into a supervised environment for 24-hours arriving no later than 0730. Blood draws will then be taken every 4 hours (0800, 1200, 1600, 2000, 2400 and 0400). Care will be taken to ensure the total blood draws (including the screening visit) stay within Red Cross Guidelines (less than 500 ml every 8 weeks).
  Groups: Cohort 1: Diurnal Variation Group
Other: External Stress Group — 2 visits will be required, each lasting approximately 2.5 hours in the afternoon.
  At both visits participants will rest quietly for 15 minutes, then have 3 blood draws and 4 saliva samples over approximately one hour. Participants will also be required to complete short questionnaires about their mood and experience.
  At the second visit, participants will also complete some thinking and talking tasks. In addition the autonomic nervous system of the participant's will be monitored throughout the visit.
  Groups: Cohort 2: External Stress Group

SUMMARY:
Despite advances in AntiRetroviral Therapy (ART) leading to a rapid control of the HIV virus in individuals affected, HIV can persist indefinitely and there is no cure. The HIV virus has been shown to have a unique ability to hide within the human gene inside human cells and in tissues, remaining 'silent' and rapidly reactivate 'waking up" if ART is stopped.

There are a number of ways to measure the silent HIV reservoir, including a common research-based laboratory test called Cell-Associated UnSpliced (CA-US) HIV RNA. This is an early marker of the HIV virus waking up. It is often used to test how well new drugs developed to eliminate the silent virus might work.

This study is examining whether the diurnal variation (daily rhythm) and/or stress can affect CA-US HIV RNA levels in individuals diagnosed with HIV and receiving ART.

DETAILED DESCRIPTION:
Undetectable or low circulating levels of HIV virus in blood are the result of people who have been diagnosed with a HIV-infection and who have adhered to a HIV AntiRetroviral Therapy (ART) regimen. However, the ART has not eradicated the virus from the body and individuals who cease ART can rapidly revert from a well-controlled state to showing high levels of HIV virus in the blood. The HIV virus has been shown to have a unique ability to hide within the human gene inside human cells and in tissues, remaining 'silent' and rapidly reactivate [or wake up] if ART is stopped. Efforts are underway to explore novel ways to entirely eradicate HIV from individuals, so that people who are HIV-infected can stop treatment and still have undetectable HIV viral load and remain well despite not being on HIV treatment.

There are a number of ways to measure the silent HIV reservoir, including a common research-based laboratory test called Cell-Associated UnSpliced (CA-US) HIV RNA. This is an early marker of the HIV virus reactivating. It is often used to test how well new drugs developed to eliminate the silent virus might work.

Recently as investigators involved in another clinical study, an unexpected observation was noted in a group of HIV study participants on ART between the CA-US HIV RNA levels and time of blood collection. Levels of CA-US HIV RNA appeared to be lower when blood samples were collected earlier in the morning. However, at the time of this observation, as investigators were unable to establish whether this discrepancy could be due to (i) the diurnal variation or (ii) unknown stress factors that may have been experienced by the study participants. It has previously been demonstrated that individuals with untreated HIV infection there is a variation in HIV RNA levels and the time of day. However, the effects of external factors such as time of day or stresses on CA-US HIV RNA levels in individuals while on ART have not been previously examined.

This study hopes to explore and answer the questions (i) Does the diurnal variation play a role in regulating the levels of CA-US HIV RNA in blood of individuals diagnosed with HIV and receiving ART and (ii) Does stress affect the levels of CA-US HIV RNA.

Understanding some factors that affect levels of CA-US HIV RNA may provide a new perspective on ways to eliminate the silent virus.

ELIGIBILITY:
Inclusion Criteria:

* Male
* HIV +
* On suppressive ART > 3 years
* Undetectable viral load, documented in past 3 months
* English speaking
* Have regular sleeping habits (~ 6 - 8 hours a night) [Cohort 1]
* Do not do shift-work [Cohort 1]
* Have not had any transcontinental travel in the last month [Cohort 1]

Exclusion Criteria:

* Known sleep disorder, Addison's disease, diabetes or thyroid/pituitary/adrenal/splenic disorder (note: corrected hypothyroid disorder may be allowed if recent Thyroid Stimulating Hormone (TSH) results are within normal limits);
* Current cancer (radiation, chemo or surgery within past year);
* Recent anemia
* Medications that affect study outcomes, including Automatic Nervous System (ANS) measurement: Use of immunomodulation drugs (e.g. Interleukin 21, prednisone, growth hormone, tacrolimus, methotrexate; or other medications used in autoimmune disorders such as lupus, rheumatoid arthritis, Crohn's disease, MS)
* Steroids including; corticosteroids (including regular use of inhaled/nasal steroids for severe/chronic asthma or allergies), testosterone, or anabolic steroids
* Beta-blockers
* Certain psychiatric medications including regular use of medium or long-acting benzodiazepines or other anxiolytics/sedatives (note: occasional use of short-acting anxiolytics or sleep meds okay);
* Disulfiram or experimental Latent Retroviral Activation (LRA) use
* Psychiatric conditions including current major depression or severe anxiety disorder; bipolar disorder; schizophrenia; current PTSD; or severe Attention Deficit Hyperactivity Disorder (ADHD)
* Alcohol use > 14 drinks/week, or daily use of any recreational drug other than marijuana (participant must be able abstain from alcohol and recreational drug use the day before and day of study visits)
* BMI>34.9
* Pacemaker
* General anesthesia in the past month
* Inability to provide informed consent

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cohort 1: Open to study participants who meet the inclusion/exclusion criteria and have been either referred by their health care provider or self-referred to the study team.
  Cohort 2: Open to study participants who meet the inclusion/exclusion criteria; participants will be primarily drawn from the pool of Options and Scope study participants who have consented to being contacted for future studies
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Diurnal variation effects on HIV transcription | 24 hours
  To determine if there are diurnal variations in cortisol and catecholamine in HIV transcription in latently-infected cells in HIV-infected participants on ART.
Stress Factor effects on HIV transcription | Baseline (visit 1) and visit 2 (approximately 1 - 7 days later)
  To determine the effects of stress-induced changes in cortisol and catecholamine on HIV transcription, in latently infected cells in HIV-infected participants on ART.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon R Lewin, FRACP, PhD, Principal Investigator — The Doherty Institute for Infection and Immunity, Melbourne University; Frederick M Hecht, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Osher Center, University of California San Francisco, San Francisco, California
  - Division of Infectious Diseases, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No